CLINICAL TRIAL: NCT05358327
Title: Safety and Efficacy of Sofwave Treatment to Lift Upper Arm Lax Skin
Brief Title: Treatment for Lifting Upper Arm Lax Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sofwave Medical LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sofwave07
Record Dates: First submitted 2022-04-19; First posted 2022-05-03 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2022-03

CONDITIONS: Lax Skin
Keywords: upper arms, lax skin
MeSH Terms: conditions — Cutis Laxa; Rhabdomyosarcoma, Alveolar

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Upper Arm (Experimental)
  Interventions: Device: Sofwave

INTERVENTIONS:
Device: Sofwave — The Sofwave System, comprised of an applicator and a console, generates high intensity, non-focused ultrasonic energy which can be delivered percutaneously to tissues.
  Other Names: SUPERB

SUMMARY:
Open-label, non-randomized, prospective, multi-center, self-controlled clinical study with masked evaluation.

DETAILED DESCRIPTION:
Eligible patients will receive 2 treatments on both upper arms (4-6 weeks apart) using the Sofwave System.

Treatment may be administered after the enrollment and screening at the first visit, or it may occur later following the enrollment and screening activities based on site scheduling availabilities. All patients will return to the clinic for follow up visit at 3 months ± 2 weeks post last treatment (FU1).

Methodology described in the protocol to evaluate efficacy and safety of treatments will be carried out at each visit at the clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects > 35 years of age and < 70 years of age.
2. Not pregnant or lactating and must be either post-menopausal, surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment (i.e., oral contraceptives, contraceptive implant, barrier methods with spermicide) or abstinence.
3. Desire to undergo upper arms skin lax lifting treatments.
4. Subject has clearly visible lax skin on the upper arm, which in the investigator's opinion, may benefit from the treatment.
5. Subject agrees to maintain his/her weight (i.e., within 5% of total body weight) by not making any major changes in their diet or exercise routine during the course of the study.
6. Able and willing to comply with all visits, treatments and evaluations schedules and requirements.
7. Willing to have research photos taken of treatment areas.
8. Subject agrees not to undergo any other upper arm skin lax treatments for a period of 3 months following Sofwave treatment.
9. Able to understand and provide written Informed Consent.

Exclusion Criteria:

1. Pregnant or planning to become pregnant, having given birth less than 3 months ago, and/or breast feeding.
2. Skin disorders (skin infections or rashes, extensive scarring, psoriasis, etc.) in the treatment area.
3. Medical disorder that would hinder the wound healing or immune response (such as blood disorder, inflammatory disease, etc.).
4. History of Epileptic seizures.
5. Known allergy to lidocaine or epinephrine or antibiotics.
6. Active malignancy or history of malignancy in the past 5 years.
7. Suffering from significant concurrent illness, such as cardiac disorders, diabetes (type I or II), lupus, porphyria, or pertinent neurological disorders (i.e. any disease state that in the opinion of the investigator may interfere with the anesthesia, treatment, or healing process).
8. History of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications.
9. Suffering from hormonal imbalance, whether related to thyroid, pituitary, or androgen.
10. History of significant lymphatic drainage problems.
11. Currently heavy smoker or has history of heavy smoking (25 cigarettes per day or more) in past 10 years.
12. History of chronic drug or alcohol abuse.
13. History of bleeding disorder or is taking any medication that in the investigator's opinion may increase the subject's risk of bruising.
14. Currently taking or has taken diet pills or weight control supplements within the past month.
15. BMI>=30kg/m2
16. Non-stable weight nominally ±5% for at the past month.
17. Active implanted device such as a pacemaker, defibrillator, or drug delivery system.
18. History of epidermal or dermal disorders (particularly involving collagen or microvascularity), including collagen vascular disease or vasculitic disorders.
19. History of a fat reduction procedure (e.g., liposuction, surgery, lipolytic agents, etc.).
20. History of prior surgery in the upper arms.
21. Excessive subcutaneous fat on the upper arms.
22. Severe solar elastosis on the intended to treat area.
23. Significant scarring, atrophic scars in the area to be treated, or has a history of atrophic scars or keloids or prone to bruising.
24. Tattoo or former tattoo at or near treatment area.
25. Presence of an implant in or adjacent to area of intended treatment (upper arms).
26. History of ablative or non-ablative resurfacing/rejuvenation laser treatment or light treatment within the past 6 months, dermabrasion or deep peeling within the past 12 months on the intended to treat area.
27. Inability to understand the protocol or to give informed consent.
28. On-going use of psychiatric medication.
29. Unable or unwilling to comply with the study requirements and procedures.
30. Currently enrolled in a clinical study of any other unapproved investigational drug or device.
31. Any other condition that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Rate of improvement of upper arms lax skin | 1 year
  following Sofwave treatment as evaluated by independent masked reviewers

CONTACTS AND LOCATIONS:
Overall Officials: Ruthie Amir, MD, Study Director — CMO
Locations (4):
- United States (4):
  - Laser & Skin Surgery Center of Northern California, Sacramento, California
  - Advanced Dermatology, Lincolnshire, Illinois
  - Laser & Skin Surgery Center of New York®, New York, New York
  - Main Line Center for Laser Surgery, Ardmore, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided